CLINICAL TRIAL: NCT06981793
Title: Predictors of Anesthesia Complications in Patients Undergoing Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Gonesse (Other)
Responsible Party: Sponsor
Other Study IDs: 0050_ANESTHESIE
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Bariatric Surgery; Anesthesia, General; Postoperative Complications; Obesity; Risk Factors
MeSH Terms: conditions — Postoperative Complications; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to identify factors that can predict complications related to anesthesia in patients undergoing weight-loss surgery. By looking at patient data from past surgeries, we hope to better understand which factors increase the risk of anesthesia problems, helping doctors improve patient safety during these procedures.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥ 18 years)
* Patients who underwent a longitudinal gastrectomy (sleeve) between January 1, 2020, and June 30, 2021, at CHG, as part of bariatric surgery treatment.

Exclusion Criteria:

* Minor patients
* Patients who underwent a bariatric surgery other than sleeve gastrectomy
* Patients who objected to the use of their data for research purposes

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study participants will be selected from adult patients who underwent sleeve gastrectomy as part of bariatric surgery at the Gonesse Hospital (CHG) between January 1, 2020, and June 30, 2021.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
Occurrence of Anesthesia-Related Complications in Bariatric Surgery Patients | October 2023 - January 2024
  The primary outcome of this study is to assess the occurrence of anesthesia-related complications in patients undergoing bariatric surgery, specifically sleeve gastrectomy. These complications include difficult intubation, bronchospasm, desaturation, abnormal heart rate (bradycardia or tachycardia), changes in blood pressure (hypotension or hypertension), nausea and vomiting, hypo or hyperglycemia, delayed awakening, and death. This measure will help identify factors that predict the likelihood of these complications, ultimately improving patient safety in bariatric surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- France, Gonesse, France, France